CLINICAL TRIAL: NCT06406556
Title: Evaluate the Safety and Efficacy of Pegaspargase-based Concurrent Chemoradiotherapy in the Treatment of Early Stage Extranodal NK/T Cell Lymphoma
Brief Title: Safety & Efficacy of Peg-ASP-based CCRT in Early Stage ENKTL
Acronym: ENKTL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hua Wang, Associate senior doctor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2018-053
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Extranodal NK/T-cell Lymphoma
Keywords: extranodal NK/T-cell lymphoma; concurrent chemoradiotherapy; pegaspargase
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell

STUDY DESIGN:
Intervention Model Description: Patients receive CCRT (radiation 50 Gy and two cycles of pegaspargase 2500 unit/m2 every 3 weeks) followed by 4 courses of pegaspargase.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients diagnosed with early ENKTL. (Experimental): Patients received 4 cycles of pegaspargase including CCRT ( involved field radiotherapy 50GY, concurrent 2 cycles of pegaspargase treatment ).
  Interventions: Combination Product: Pegaspargase combined with concurrent radiotherapy.

INTERVENTIONS:
Combination Product: Pegaspargase combined with concurrent radiotherapy. — Patients receive CCRT (radiation 50 Gy and two cycles of pegaspargase 2500 unit/m2 every 3 weeks). 4 courses of pegaspargase were performed after CCRT.

SUMMARY:
The purpose of this multi-center, single arm, phase Ⅱ clinical trail is to evaluate the efficacy and toxicity of concurrent chemoradiotherapy by using single-drug pegaspargase for patients with ENKTL in stage IE to IIE.

DETAILED DESCRIPTION:
The treatment regimen included CCRT ( involved field radiotherapy 50GY, concurrent 2 cycles of pegaspargase treatment ) followed by 4 cycles of pegaspargase. Chemotherapy and RT were performed simultaneously within one week after enrollment. The administration regimen was as follows : day1, deep intramuscular injection of 2500 unit/m2 pegaspargase at three different sites, and repeated once every 3 weeks. 3D conformal radiotherapy was performed using 4 or 6 MV photons generated by a linear accelerator. The radiation dose was 50 Gy, 2.0 Gy / time, 1 time / d, for 5 weeks. The clinical target volume ( CTV ) of limited stage IE patients was defined as bilateral nasal cavity, bilateral ethmoid sinus and ipsilateral maxillary sinus. The CTV of extensive stage IE patients was extended to the affected tissues. The CTV of stage IIE lesions also included the involved cervical lymph node area.

ELIGIBILITY:
Inclusion Criteria:

1.The patient was pathologically diagnosed as ENKTL and had not received any previous treatment for ENKTL;2.The estimated survival time ≥ 3 months. 3.18-75 years old ; 4. Ann-Arbor stage was IE-IIE ; 5. ECOG performance status 0-2 ; 6.Clinicians judged that patients were suitable for concurrent chemoradiotherapy ; 7.No radiotherapy or hormone drugs were received within 4 weeks before treatment;8.After the patients were enrolled in the trial, they could not accept other drugs that may have therapeutic effects on ENKTL ; 9.WBC≥ 3 × 109 / L, NE ≥ 1.5 × 109 / L, PLT ≥ 100 × 109 / L ; 10.Serum creatinine ≤ 1.5mg / dL, creatinine clearance rate ≥ 50mL / min ; 11.ALT, AST ≤ 3 × ULN ( normal upper limit ) ; total bilirubin ≤ 2 × ULN ; 12.Serum fibrinogen level ≥ 1.0g / L ; 13.Signed informed consent form.

Exclusion Criteria:1.Symptomatic CNS involvement, previous or current accompanied by other malignant tumors ; 2.The primary lesion is ENKTL from non-upper respiratory gastrointestinal tract ; 3.Patients with poor general condition, ECOG performance status >2 ; 4.Women in pregnancy or lactation; 5.The patient ( male or female ) has the possibility of fertility but is unwilling or does not take effective contraceptive measures; 6. Known allergies to test drugs or any excipient component of these products ;7.Doctors believe that patients are not suitable for concurrent chemoradiotherapy; 8.Active infection ( determined by the researcher ) ; 9.According to the researchers ' judgment, there are concomitant diseases that seriously endanger the safety of patients or affect the completion of the study;10. Have a clear history of neurological or psychiatric disorders, including epilepsy or dementia.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2016-03-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
PFS | From enrollment to the end of treatment at 2 years
  progression free survival (PFS) rate

SECONDARY OUTCOMES:
OS | From enrollment to the end of treatment at 2 years
  two-year overall survival rate
CRR | From enrollment to the end of treatment at 2 weeks
  complete response rate

CONTACTS AND LOCATIONS:
Overall Officials: Hua Wang, MD, Principal Investigator — Sun Yat-senU
Locations (1):
- HuaWang, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No